CLINICAL TRIAL: NCT07405320
Title: Testing a Brief Video Intervention to Support Patient Coping Following Radioiodine Treatment
Brief Title: A Brief Video Intervention to Improve Patient Outcomes Following Radioiodine Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Keith J Petrie, Principal Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24301
Record Dates: First submitted 2025-11-18; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Thyroid Cancer; Hyperthyroidism; Radioiodine Treatment
Keywords: Mindset; Digital Intervention; Radioiodine
MeSH Terms: conditions — Thyroid Neoplasms; Hyperthyroidism

STUDY DESIGN:
Intervention Model Description: This study is a two-arm parallel randomised controlled trial. Prior to treatment, participants will be randomly assigned to one of two arms. The control group will view a neutral video that discusses general health advice unrelated to the radioiodine treatment, while the intervention group will view a video that reframes side effects and safety instructions in a more adaptive way. Outcomes will then be compared between the two groups in terms of side effects, disability and understanding of treatment precautions.
Who Masked: Participant
Masking Description: To control for expectation effects both groups will be told that we are testing different videos to assist patients with the radioiodine treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Video (Experimental): Participants assigned to the intervention group will view a brief video that explains radioiodine treatment, side effects, and radiation safety requirements using adaptive and supportive framing.
  Interventions: Behavioral: Intervention Video
- Control Video (Active Comparator): Participants assigned to the control group will view a neutral video containing general health-related information unrelated to radioiodine treatment. The video will be similar in length, style, and presenter to the intervention video.
  Interventions: Behavioral: Control Video

INTERVENTIONS:
Behavioral: Intervention Video — Participants will view a brief prerecorded video (approximately 4 minutes) online, delivered through Qualtrics, following completion of the baseline questionnaire. The intervention video will present information on radioiodine treatment recovery, managing treatment side effects, and radiation safety requirements. The video will be delivered online prior to the participant's radioiodine treatment, using patient-friendly language and supportive framing.
  Arms: Intervention Video
Behavioral: Control Video — Participants will view a brief prerecorded neutral video (approximately 4 minutes) online, being delivered through Qualtrics following the baseline questionnaire. The control video will present general health information unrelated to radioiodine treatment (e.g., healthy lifestyle topics such as nutrition and stress management). The video will be delivered online prior to the participant's radioiodine treatment, and will match the intervention video in duration, format, and presenter.
  Arms: Control Video

SUMMARY:
This study will test the impact of a short video intervention for people who are receiving radioiodine treatment for thyroid conditions (such as hyperthyroidism or thyroid cancer). After their single-dose treatment, patients need to follow safety instructions to protect others and manage side effects during recovery. Some people find these instructions hard to remember, and side effects (or anticipation of side effects) can feel worrying or disruptive. The video aims to present the treatment information in a more accessible patient-friendly way, so that patients feel less distressed, find their side effects easier to cope with, and better engage with safety precautions. All patients will first have a pre-treatment consultation with their doctor and receive the standard treatment information currently provided. Before this consultation patients will be randomly assigned to view one of two videos. The control group will see a neutral video that details standard health information that is not specific to radioiodine, while the intervention group will see a video that explains side effects, safety requirements and recovery period in a more adaptive way. Comparing these two groups will allow us to assess whether this new approach improves coping, reduces distress, and enhances adherence to safety instructions in the post-dose recovery phase of radioiodine treatment.

DETAILED DESCRIPTION:
This study is a two-arm randomised controlled trial. Prior to treatment, participants will be randomly assigned to one of two arms. The control group will view a neutral video that discusses general health advice unrelated to the radioiodine treatment, while the intervention group will view a video that reframes side effects and safety instructions in a more adaptive way. All participants will receive a standard pre-treatment consultation with their doctor and the usual written information. Outcomes will then be compared between the two groups in terms of side effects, disability and understanding of treatment precautions. To control for expectation effects both groups will be told that we are testing different videos to assist patients with the radioiodine treatment. This study aims to find out whether a short video intervention (1) helps patients cope better with side effects and get back to normal activities more quickly, (2) improves how well patients remember and understand the safety instructions they need to follow after their dose, (3) reduces disability related to the treatment and its side effects. By examining whether a brief video intervention improves coping with side effects, understanding of safety instructions, and post-treatment recovery, the research will provide new knowledge on how information about radioiodine can be delivered more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Clinical diagnosis of hyperthyroidism or thyroid cancer
* Scheduled to receive radioiodine therapy at Auckland City Hospital Radiation Oncology Clinic
* Able to understand and communicate in English
* Access to an internet-connected device to complete study questionnaires

Exclusion Criteria:

* Completed previous radioiodine treatment
* Self-reported difficulty completing questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Post-treatment functional Interference | From treatment to post-treatment questionnaire (on the last day of radiation safety requirements; approximately 5-7 days post-dose) and at 4-week follow-up.
  Patient-reported functional interference following radioiodine treatment, assessed using a Functional Interference Questionnaire adapted from standard symptom interference measures. Participants rate the extent to which treatment-related effects interfere with daily activities including work, household tasks, and social participation. Each item is rated on a numeric rating scale from 0 to 10, where 0 = No interference, and 10 = Complete interference (i.e., higher scores indicate worse functioning or greater interference). A mean functional interference score will be calculated across items.
Symptom Attribution to Treatment | Pre-dose (1-3 weeks prior to treatment), post-dose (approximately 5-7 days post-dose), and 4-week follow-up.
  Symptom attribution assessed using the Side Effect Attribution Scale (SEAS), which measures the extent to which participants attribute experienced symptoms to radioiodine treatment rather than to other causes. Participants rate attribution for 52 symptoms using a a 5-point Likert scale (i.e., 1-5 range):
  1. = Definitely not a side effect
  2. = Probably not a side effect
  3. = Unsure
  4. = Probably a side effect
  5. = Definitely a side effect Higher scores indicate greater attribution of symptoms to treatment, whilst scores near 3 indicate uncertainty. A total attribution score is calculated by averaging responses across all symptoms.
Adherence to Radiation Safety Precautionary Behaviours | From treatment to post-treatment questionnaire (on the last day of radiation safety requirements; approximately 5-7 days post-dose) and at 4-week follow-up.
  Self-reported adherence to recommended radioiodine radiation safety precautionary behaviours (e.g., distancing, hygiene practices), assessed using a structured adherence questionnaire developed for this study.
  Adherence is quantified as a composite adherence score, calculated as the proportion of prescribed precautionary behaviours adhered to, with values ranging from 0 to 100%, where higher scores indicate greater adherence.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including item-level questionnaire responses and derived summary scores collected at each study time point (e.g., symptom attribution scores, functional interference scores, and adherence scores), as well as basic demographic variables necessary to reproduce the primary analyses.
  Data that could directly or indirectly identify individual participants (e.g., names, contact details, dates of birth) will not be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The start date will be after publication of the primary results or completion of the thesis, whichever occurs first. IPD will be available upon reasonable request for up to 5 years following study completion.
Access Criteria: De-identified IPD and supporting information will be available to qualified researchers upon reasonable request. Requests must include a brief proposal outlining the intended use of the data and will be reviewed by the study investigators. Approved requestors will be granted access to de-identified datasets and supporting documentation via secure data transfer. Data sharing will be conducted in accordance with institutional ethics approval and data governance requirements.